CLINICAL TRIAL: NCT05060705
Title: Randomized Controlled Open Study of Safety and Preliminary Efficiency of the Drug "Efesovir" (Oral Solution) for Coronavirus Infection (COVID-19)
Brief Title: "Efesovir" (FS-1) for COVID-19, Phase 2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scientific Center for Anti-infectious Drugs, Kazakhstan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-FS-1-SE-2-05
Record Dates: First submitted 2021-09-24; First posted 2021-09-29 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: COVID19; viral pneumonia; FS-1; Efesovir
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — pharmaceutical FS-1

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the one of two parallel groups: 1) treated with study drug "Efesovir"; 2) treated with referent drug "Remdesivir".
Masking Description: no masking, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efesovir (Experimental): The patients of experimental arm take study drug Efesovir twice a day as an antiviral therapy in dose 0.125 ml / kg. Daily dose of Efesovir: 0.250 ml / kg. Duration of treatment is 5 - 10 days, depending on the severity of the disease.
  Interventions: Drug: Efesovir
- Remdesivir (Active Comparator): The patients are treated with the antiviral drug "Remdesivir" in dose 200 mg intravenously on the 1st day, then by 100 mg intravenously daily for 5 - 10 days, depending on the severity of the disease.
  Interventions: Drug: Efesovir

INTERVENTIONS:
Drug: Efesovir — Antiviral therapy of COVID19 with Efesovir oral solution in dose 0.125 ml / kg two times per day. Duration of treatment is 5 - 10 days, depending on the severity of the disease.
  Other Names: FS-1

SUMMARY:
Study of the efficacy and safety of the new drug "Efesovir" in comparison with the drug "Remdesivir" in the treatment of patients hospitalized with COVID-19.

The hypothesis of clinical study is the clinical efficacy of new drug "Efesovir" is 10% to 30% higher than of "Remdesivir".

ELIGIBILITY:
Inclusion Criteria:

* polymerase chain reaction (PCR) confirmed coronavirus infection (COVID-19) in hospitalized patients with severe risk factors in age from 18 years to 59 years, of both sexes, irrespective of national or ethnic origin
* the duration of the COVID-19 disease is no more than 10 days
* informed concent to participate in clinical trials
* informed concent to to use reliable contraceptive methods while participating in a clinical trial

Exclusion Criteria:

* age less than 18 years old and over 59 years old
* pregnancy or breastfeeding
* hypersensitivity, allergy, intolerance to iodine, iodine-containing medicines
* hypersensitivity to Remdesivir or its components
* impaired consciousness, causing the impossibility of oral administration
* conditions or circumstances that, in the opinion of the investigator, may affect the patient's safety or the quality of the results obtained
* participation in another clinical trial, including in the period up to 2 months before this study
* signs of multiple organ failure
* alanine aminotransferase (ALT), aspartate aminotransferase (AST) is 5 or more times higher than normal
* thrombocytopenia below 100 * 10^9/ l
* decrease in glomerular filtration rate (GFR) less than 30 ml / min by 1.73 m2
* chronic heart failure with reduced ejection fraction
* liver failure
* coagulopathy
* mechanical ventilation for 48 hours or more
* extracorporeal membrane oxygenation (ECMO)
* disseminated intravascular coagulation

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Response Rate | 21 days
  Clinical Response Rate is calculated as the number of trial subjects with effective treatment over the total number of subjects multiplied by 100. It is calculated in each study group.
  Measured in percents. The outcome is estimated among randomized subjects completed clinical study with the protocol requirements (per protocol population (PPP)).
  Clinical response is evaluated as effective treatment if: all signs and symptoms of COVID19 are resolved or improved with no worsening or appearance of new signs and symptoms; there is no requirement for additional antiviral of antibacterial therapy; chest roentgenograms (CT scans) are improved. The outcome is assessed in day 21 from the start of Study Drug treatment (visits 13).

SECONDARY OUTCOMES:
Early Clinical Response Rate | 72 hours (3 days) of study drug treatment
  Early clinical response rate defined as complete resolution or significant improvement of at least 2 of 4 leading baseline signs and symptoms within 72 hours after the start of Study (Referent) Drug treatment. It is estimated in the Intent to Treat (ITT) population. The outcome is measured in percents.
Early Clinical Response Rate in pneumonia | 72 hours (3 days) of study drug treatment
  The outcome is estimated in patients with pneumonia due to coronavirus infection (modified ITT population). It is defined as complete resolution or significant improvement of at least 2 of 4 main clinical symptoms of pneumonia (cough, shortness of breath, chest pain, sputum) within 72 hours after the start of Study (or Referent) Drug treatment. The outcome is measured in percents. The percentage of subjects with an early clinical response to pneumonia in the compared groups is statistically estimated.
Percentage of clinically stable patients | 72 hours (3 days) of study drug treatment
  Percentage of patients at Day 3 who are clinically stable.
  Clinical stability defined as:
  * Blood oxygen saturation >= 93%
  * Temperature <=38.0°C
  * Heart rate <=100 beats per minute
  * Respiratory rate <=25 per minute
  * Systolic blood pressure ≥90 mm Hg
  * Ability to maintain oral intake
  * Normal mental status (oriented to person, place or time) A patient is considered to be clinically stable if all stability criteria are met. The outcome is assessed in ITT population. The difference between groups in the percentage of clinically stable patients from the total number of study subjects in the group is statistically evaluated.
Survival rate | 21 days
  Percentage of participants surviving at day 21. The indicator is calculated as the number of live subjects at the last visit (day 21) divided by the total number of study subjects in the group multiplied by 100.
  The outcome is estimated among subjects who completed the study in compliance with the protocol (per protocol population (PPP)).
Clinical Status Change | 7 days
  The clinical status is determined by the ordinal scale:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities and/or requiring home oxygen
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care
  5. Hospitalized, requiring supplemental oxygen
  6. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  7. Hospitalized, on invasive mechanical ventilation or Extracorporeal Membrane Oxygenation
  8. Death
  Clinical status is assessed in ITT population. The outcome is recorded at all visits, starting from the day of randomization. A decrease in points indicates the effectiveness of treatment. When the indicator changes during the day, the worst score of the day is recorded. Statistical analysis is performed on the Day 7 from the start Study Drug treatment, comparing with the score at randomization.
Adverse Events (AE) | up to 21 days
  The safety of Study Drug (Referent Drug) will be assessed by adverse event and serious adverse event monitoring.
Thyroid gland function | Day 21
  Changes in laboratory parameters of thyroid gland function (hormones) at the last visit in comparison with the baseline data (thyroid stimulating hormone (TSH), free triiodothyronine (FT3)).

CONTACTS AND LOCATIONS:
Locations (1):
- Semey Medical University, Semey, East Kazakhstan, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
all individual participant Data (IPD )that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2022
Access Criteria: written request
URL: http://scaid.kz/

REFERENCES:
- See also: Yuldasheva, G., R. Argirova and A. Ilin. "A quantum-chemical model of the inhibition HIV-1 integrase action by iodine complex compounds and lithium halogenides." Journal of AIDS and Clinical Research 6 (2015): 1-6. DOI:10.4172/2155-6113.1000465 Corpus — http://www.hilarispublisher.com/open-access/a-quantumchemical-model-of-the-inhibition-hiv1-intergrase-action-by-iodine-complex-compounds-and-lithium-halogenides-2155-6113-1000465.pdf
- See also: Yuldasheva, G. , Zhidomirov, G. and Ilin, A. (2011) A quantum-chemical model of the inhibition mechanism of viral DNA HIV-1 replication by Iodine complexcompounds. Natural Science, 3, 573-579. doi: 10.4236/ns.2011.37080 — http://www.scirp.org/html/6374.html
- Available data/document: thesis of online seminar — http://infectiousdiseases.heraldmeetings.com/0 — Gulnara A Yuldasheva and A I Ilin Inhibition of the catalytic fragment of the ExoN domain of the exoribonuclease of SARS-CoV-2-betacoronavirus B virus by FS-1 drug containing molecular iodine and lithium and magnesium halides International conference on infectious diseases, Infectious Diseases Prevention, Control and Cure, August 27 - 28, 2020 online seminar